CLINICAL TRIAL: NCT00681928
Title: The Effect of Aromatase Inhibition on the Cognitive Function of Older Patients With Breast Cancer
Brief Title: Cognitive Function in Older Women With Stage I, Stage II, or Stage III Breast Cancer Receiving Hormone Therapy
Status: Completed | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 07006; P30CA033572 (NIH); CHNMC-07006; CDR0000589001 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2008-05-20; First posted 2008-05-21 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-11

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Letrozole; Mental Status and Dementia Tests; Psychiatric Rehabilitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Breast Cancer patients receiving aromatase treatment
  Interventions: Drug: anastrozole; Drug: letrozole; Other: questionnaire administration; Procedure: cognitive assessment; Procedure: psychosocial assessment and care
- Healthy female controls age 60 and older
  Interventions: Other: questionnaire administration; Procedure: cognitive assessment; Procedure: psychosocial assessment and care

INTERVENTIONS:
Drug: anastrozole — As determined by the subject's physician
  Groups: Breast Cancer patients receiving aromatase treatment
Drug: letrozole — As determined by the subject's physician
  Groups: Breast Cancer patients receiving aromatase treatment
Other: questionnaire administration — For cancer patients prior to starting medication and 6 months after starting medication. For healthy controls, one time administration.
Procedure: cognitive assessment — For cancer patients prior to starting medication and 6 months after starting medication. For healthy controls, one time administration.
Procedure: psychosocial assessment and care — For cancer patients prior to starting medication and 6 months after starting medication. For healthy controls, one time administration.

SUMMARY:
RATIONALE: Gathering information about cognitive function over time in postmenopausal women with breast cancer may help doctors learn about the long-term effects of aromatase inhibitor therapy and plan the best treatment.

PURPOSE: This clinical trial is studying cognitive function in older postmenopausal women with stage I, stage II, or stage III breast cancer receiving hormone therapy and in healthy volunteers.

DETAILED DESCRIPTION:
OBJECTIVES:

* Explore the impact of treatment with an aromatase inhibitor on the cognitive function of postmenopausal women with stage I-III breast cancer vs in cancer-free, age-matched healthy volunteers.

OUTLINE: Patients receive adjuvant anastrozole or letrozole in the absence of disease progression or unacceptable toxicity.

Patients and healthy volunteers undergo cognitive function testing consisting of neuropsychological battery tests and complete self-reported questionnaires (e.g., Squire Memory Self-Rating Questionnaire, and FACT-B Quality of Life Measure) regarding cognitive ability, quality of life, fatigue, and psychosocial status. Patients and healthy volunteers also undergo geriatric assessment at baseline and after 6 months of initiation with aromatase inhibitor therapy.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Patient diagnosed with breast cancer

    * Stage I-III disease
    * Estrogen receptor- and/or progesterone receptor-positive
    * Planning to start treatment with anastrozole or letrozole
  * Age-matched healthy volunteer (control)

    * No history of breast cancer
    * Not receiving adjuvant aromatase inhibitor therapy

PATIENT CHARACTERISTICS:

* Postmenopausal
* Able to converse, write, and read English
* No claustrophobia (patients participating in the PET scan correlative study)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior hormonal therapy, including estrogen replacement therapy
* No previous treatment with CNS radiation

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Breast cancer patients and healthy control subjects
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2007-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Impact of treatment with an aromatase inhibitor on cognitive function | Prior to starting aromatase treatment and 6 months after starting the medication.

CONTACTS AND LOCATIONS:
Overall Officials: Arti Hurria, MD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States

REFERENCES:
- [Derived] Hurria A, Patel SK, Mortimer J, Luu T, Somlo G, Katheria V, Ramani R, Hansen K, Feng T, Chuang C, Geist CL, Silverman DH. The effect of aromatase inhibition on the cognitive function of older patients with breast cancer. Clin Breast Cancer. 2014 Apr;14(2):132-40. doi: 10.1016/j.clbc.2013.10.010. Epub 2013 Oct 25. PMID 24291380